CLINICAL TRIAL: NCT05798845
Title: Exploratory Phase II Clinical Study of Toripalimab Plus Radiotherapy Versus Toripalimab Plus Chemotherapy for the Neoadjuvant Treatment of Operable Stage II-IIIA (N+) Non-small Cell Lung Cancer (NSCLC)
Brief Title: The Effect of Toripalimab Plus Radiotherapy in Patients With Operable Stage II-IIIA (N+) Non Small Cell Lung Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Chest Hospital (Other)
Collaborators: Shanghai Junshi Bioscience Co., Ltd. (Other)
Responsible Party: Principal Investigator, Xiaolong Fu, director,department of radiation oncology, Shanghai Chest Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: neoRT-Lung
Record Dates: First submitted 2023-01-18; First posted 2023-04-05 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: NSCLC
Keywords: neoadjuvant immunotherapy; radiotherapy
MeSH Terms: interventions — toripalimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A (Experimental): Radiation: primary tumor SBRT, DT: 24Gy/3Fx, d1-3; positive lymph nodes LDRT, DT: 2Gy/2Fx, d1-2, d22-23 (2 cycles) ; Drug: toripalimab 240mg ivgtt d4, d24 (2 cycles)
  Interventions: Radiation: SBRT+LDRT; Drug: Toripalimab
- Arm B (Active Comparator): Drug: Chemotherapy + toripalimab 240mg ivgtt d1, d22 (2 cycles)
  Chemotherapy regimen:
  Non-squamous carcinoma: pemetrexed + platinum or paclitaxel + platinum. Squamous carcinoma: paclitaxel + platinum or gemcitabine + platinum
  Interventions: Drug: Chemotherapy drug; Drug: Toripalimab

INTERVENTIONS:
Radiation: SBRT+LDRT — primary tumor SBRT, DT: 24Gy/3Fx, d1-3; positive lymph nodes LDRT, DT: 2Gy/2Fx, d1-2, d22-23 (2 cycles)
  Arms: Arm A
Drug: Toripalimab — toripalimab 240mg ivgtt d4, d24 (2 cycles)
  Arms: Arm A
Drug: Chemotherapy drug — Non-squamous carcinoma: pemetrexed + platinum or paclitaxel + platinum Squamous carcinoma: paclitaxel + platinum or gemcitabine + platinum
  Arms: Arm B
Drug: Toripalimab — toripalimab 240mg ivgtt d1, d22 (2 cycles)
  Arms: Arm B

SUMMARY:
This randomized phase II trial is to explore the clinical efficacy, safety and feasibility of neoadjuvant immunotherapy plus radiotherapy compared with neoadjuvant immunotherapy plus chemotherapy in operable stage II-IIIA (N+) non small cell lung cancer (NSCLC) and the optimal radiotherapy pattern.

DETAILED DESCRIPTION:
In recent years, the survival rate after diagnosis of non small cell lung cancer (NSCLC) has improved with advances in treatment. In terms of 5-year average overall survival (OS) by stage at the time of diagnosis, OS decreases significantly from stage IB to IIIA NSCLC, with 68% for stage IB, 53-60% for stage II, and 36% for stage IIIA. How to optimize the perioperative treatment strategy to reduce postoperative recurrence and prolong the survival of patients has raised great concern in early and mid-stage NSCLC. Radiotherapy combined with immunotherapy is suggested for advanced NSCLC in preclinical basic studies and recent clinical trials. Stereotactic body radiation therapy (SBRT) at 8 Gy × 3 Fx plays an effective immunoregulated role and can further enhance the antitumor immune response promoted by immune checkpoint inhibitors (ICIs). Although little is known about the optimal SBRT dose and fraction pattern, 6 Gy × 5 Fx or 8-9 Gy × 3 Fx have shown effectiveness in clinical studies.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 75 years old, gender is not limited.
2. ECOG performance status 0-1.
3. non-small cell lung cancer diagnosed by pathology.
4. sufficient tumor tissue available for biomarker analysis.
5. clinical staging of cT1-2N1-2M0 or T3N1M0, stage II-IIIA (8th UICC staging criteria).
6. Patients with distant metastases ruled out by CT or PET/CT and physically assessed as acceptable for radical lung cancer surgery.
7. histomolecular pathology confirming the absence of classic driver oncogene mutations in EGFR, ALK, or ROS1.
8. Basic normal function of all organs (laboratory test results within 1 week prior to enrollment).

   * Bone marrow function: absolute neutrophil count (ANC) ≥ 1.5x109 /L, platelet count ≥ 100x109 /L, hemoglobin ≥ 9g/dL.
   * Liver: serum total bilirubin ≤ 1.5 times the upper limit of normal; ALT and AST ≤ 2.5 times the upper limit of normal.
   * Kidney: blood creatinine level ≤ 1.5 times the upper limit of normal or creatinine clearance ≥ 60 ml/min and urea nitrogen ≤ 200 mg/L.
   * Urine protein <+, if urine protein + then total 24 hour protein must be <500mg.
   * Blood glucose: within normal range and/or with diabetic patients on treatment but with stable blood glucose control.
   * Pulmonary function: baseline FEV1 of at least 2L; if baseline FEV1 < 2L then FEV1 > 800ml is expected after surgery as assessed by a surgical specialist.
   * Cardiac function: no myocardial infarction within 1 year; no unstable angina; no symptomatic severe arrhythmia; no cardiac insufficiency.
9. Voluntarily participated in this study and signed the informed consent form by himself or his agent

Exclusion Criteria:

1. Pathology suggestive of compound small cell lung cancer, etc.
2. History of previous lobectomy, radiotherapy or chemotherapy.
3. Those with concurrent second primary carcinoma and a history of previous malignancy of less than 5 years (except for completely cured cervical carcinoma in situ or basal cell or squamous epithelial cell skin cancer).
4. Patients with any active autoimmune disease or a history of autoimmune disease (e.g., interstitial pneumonia, uveitis, enterocolitis, hepatitis, pituitary inflammation, vasculitis, myocarditis, nephritis, hyperthyroidism, hypothyroidism, etc.).
5. Have an active infection requiring systemic treatment or a history of active tuberculosis.
6. Known history of human immunodeficiency virus (HIV) or active chronic Hepatitis C or Hepatitis B virus infection or any uncontrolled active systemic infection requiring intravenous (iv) antimicrobial treatment.
7. Those with known presence or coexistence of other uncontrollable diseases that are not amenable to surgical treatment
8. Physical examination or clinical trial finds that, in the opinion of the investigator, may interfere with the results or place the patient at increased risk for treatment complications
9. Prior interstitial lung disease, drug-induced interstitial disease or any clinically evident active interstitial lung disease with idiopathic pulmonary fibrosis on baseline CT scan; uncontrolled massive pleural or pericardial effusion
10. Unstable systemic concomitant disease (active infection, moderate to severe chronic obstructive pulmonary disease, poorly controlled hypertensive disease, unstable angina pectoris, congestive heart failure, myocardial infarction occurring within 6 months, severe mental disorder requiring medication for control, liver, renal or other metabolic disease, neuropsychiatric pathology such as Alzheimer's disease)
11. History of congenital or acquired immunodeficiency disorders or organ transplantation
12. Received any of the following treatments:

    * Prior radiotherapy, treatment with anti PD-1, anti PD-L1 or anti PD-L2 drugs, or other drugs that synergistically inhibit T-cell receptors such as CTLA-4, OX-40, CD137.
    * Having received any investigational drug within 4 weeks
    * Concurrent enrollment in another clinical study, unless it is an observational (non-interventional) clinical study or an interventional clinical study follow-up
    * Persons who have received an antineoplastic vaccine or who have received a live vaccine within 4 weeks
    * Have undergone major surgery or had severe trauma within 4 weeks

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2025-02-20 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Pathlogical complete remission (pCR) rate | 1 year
  Pathlogical complete remission rate

SECONDARY OUTCOMES:
major pathologic response (MPR) of primary tumor | 1 year
  proportion of residual tumor ≤10%
Perioperative complications | 1 year
  complications occurring during operation
Completion of surgery | intraoperative
  whether the surgery is completed
Rate of R0 resection | 1 year
  rate of participants with tumor margin negative
treatment emergent adverse event (TEAE) | 1 year
  number of participants who have adverse events occurring during the treatment period
Event-free survival (EFS) | 3 years
  Event-free survival
Overall survival (OS) | 3 years
  Overall survival
circulating tumor DNA (ctDNA) | 1 year
  the expression of circulating tumor DNA
Immune subtypes | 1 year
  the tumor immune microenvironment subtype according to PD-L1 and tumor-infiltrating lymphocytes
PD-L1 expression | 1 year
  the status of PD-L1
Tumor mutation burden (TMB) | 1 year
  frequency of tumor gene mutation

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Chest Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Howlader N, Forjaz G, Mooradian MJ, Meza R, Kong CY, Cronin KA, Mariotto AB, Lowy DR, Feuer EJ. The Effect of Advances in Lung-Cancer Treatment on Population Mortality. N Engl J Med. 2020 Aug 13;383(7):640-649. doi: 10.1056/NEJMoa1916623. PMID 32786189
- [Background] Rami-Porta R, Bolejack V, Crowley J, Ball D, Kim J, Lyons G, Rice T, Suzuki K, Thomas CF Jr, Travis WD, Wu YL; IASLC Staging and Prognostic Factors Committee, Advisory Boards and Participating Institutions. The IASLC Lung Cancer Staging Project: Proposals for the Revisions of the T Descriptors in the Forthcoming Eighth Edition of the TNM Classification for Lung Cancer. J Thorac Oncol. 2015 Jul;10(7):990-1003. doi: 10.1097/JTO.0000000000000559. PMID 26134221
- [Background] Ko EC, Raben D, Formenti SC. The Integration of Radiotherapy with Immunotherapy for the Treatment of Non-Small Cell Lung Cancer. Clin Cancer Res. 2018 Dec 1;24(23):5792-5806. doi: 10.1158/1078-0432.CCR-17-3620. Epub 2018 Jun 26. PMID 29945993
- [Background] Wang Y, Liu ZG, Yuan H, Deng W, Li J, Huang Y, Kim BYS, Story MD, Jiang W. The Reciprocity between Radiotherapy and Cancer Immunotherapy. Clin Cancer Res. 2019 Mar 15;25(6):1709-1717. doi: 10.1158/1078-0432.CCR-18-2581. Epub 2018 Nov 9. PMID 30413527
- [Background] Demaria S, Coleman CN, Formenti SC. Radiotherapy: Changing the Game in Immunotherapy. Trends Cancer. 2016 Jun;2(6):286-294. doi: 10.1016/j.trecan.2016.05.002. PMID 27774519
- [Background] Bernstein MB, Krishnan S, Hodge JW, Chang JY. Immunotherapy and stereotactic ablative radiotherapy (ISABR): a curative approach? Nat Rev Clin Oncol. 2016 Aug;13(8):516-24. doi: 10.1038/nrclinonc.2016.30. Epub 2016 Mar 8. PMID 26951040
- [Background] Theelen WSME, Chen D, Verma V, Hobbs BP, Peulen HMU, Aerts JGJV, Bahce I, Niemeijer ALN, Chang JY, de Groot PM, Nguyen QN, Comeaux NI, Simon GR, Skoulidis F, Lin SH, He K, Patel R, Heymach J, Baas P, Welsh JW. Pembrolizumab with or without radiotherapy for metastatic non-small-cell lung cancer: a pooled analysis of two randomised trials. Lancet Respir Med. 2021 May;9(5):467-475. doi: 10.1016/S2213-2600(20)30391-X. Epub 2020 Oct 20. PMID 33096027
- [Background] Vanpouille-Box C, Alard A, Aryankalayil MJ, Sarfraz Y, Diamond JM, Schneider RJ, Inghirami G, Coleman CN, Formenti SC, Demaria S. DNA exonuclease Trex1 regulates radiotherapy-induced tumour immunogenicity. Nat Commun. 2017 Jun 9;8:15618. doi: 10.1038/ncomms15618. PMID 28598415
- [Background] Altorki NK, McGraw TE, Borczuk AC, Saxena A, Port JL, Stiles BM, Lee BE, Sanfilippo NJ, Scheff RJ, Pua BB, Gruden JF, Christos PJ, Spinelli C, Gakuria J, Uppal M, Binder B, Elemento O, Ballman KV, Formenti SC. Neoadjuvant durvalumab with or without stereotactic body radiotherapy in patients with early-stage non-small-cell lung cancer: a single-centre, randomised phase 2 trial. Lancet Oncol. 2021 Jun;22(6):824-835. doi: 10.1016/S1470-2045(21)00149-2. Epub 2021 May 18. PMID 34015311